CLINICAL TRIAL: NCT00255346
Title: Therapy of Myeloid Metaplasia-Myelofibrosis, Atypical Chronic Myeloid or Myelomonocytic Leukemia, C-Kit Positive Acute Myeloid Leukemia (AML) or High-Risk Myelodysplastic Syndrome (AML-MDS), Hypereosinophilic Syndrome, Polycythemia Vera, and Mastocytosis With Dasatinib (BMS-354825)
Brief Title: Dasatinib as Therapy for Myeloproliferative Disorders (MPDs)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0817; NCI-2012-01353 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2005-11-16; First posted 2005-11-18 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Agnogenic Myeloid Metaplasia; Myelofibrosis; Hypereosinophilic Syndrome; Polycythemia Vera; Mastocytosis; Leukemia, Myelomonocytic, Chronic
Keywords: targeted therapy; leukemia; Acute myeloid leukemia (AML); Myelodysplastic syndrome (MDS); Agnogenic myeloid metaplasia - myelofibrosis (MMM); Hypereosinophilic syndrome (HES); Polycythemia vera (PV); Mastocytosis; CMML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Primary Myelofibrosis; Hypereosinophilic Syndrome; Polycythemia Vera; Mastocytosis; Leukemia, Myelomonocytic, Chronic; Leukemia | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Acute myeloid leukemia (AML) (Experimental): Dasatinib 70 mg orally twice daily.
  Interventions: Drug: Dasatinib (BMS-354825)
- MDS/CMML (Experimental): Dasatinib 70 mg orally twice daily.
  Interventions: Drug: Dasatinib (BMS-354825)
- HES/CEL (Experimental): Dasatinib 70 mg orally twice daily.
  Interventions: Drug: Dasatinib (BMS-354825)
- Primary myelofibrosis (PMF) (Experimental): Dasatinib 70 mg orally twice daily.
  Interventions: Drug: Dasatinib (BMS-354825)
- Systemic Mastocytosis (SM) (Experimental): Dasatinib 70 mg orally twice daily.
  Interventions: Drug: Dasatinib (BMS-354825)

INTERVENTIONS:
Drug: Dasatinib (BMS-354825) — 70 mg orally twice daily
  Other Names: Sprycel

SUMMARY:
The goal of this clinical research study is to learn if dasatinib can help to control myeloproliferative disorders. The safety and tolerability of dasatinib will also be studied.

DETAILED DESCRIPTION:
Dasatinib is an experimental anti-cancer drug that is designed to block the function of BCR-ABL, which is the abnormal protein responsible for causing leukemia in some cells.

If you are found to be eligible to take part in this study, you will take dasatinib by mouth twice a day. If you have mastocytosis, you will take dasatinib by mouth once a day. A treatment cycle will be defined as 4 weeks (28 days) + 7 days. You will be instructed to take dasatinib in the morning (between about 6:00 a.m.-10:00 a.m.) and in the evening (between about 6:00 p.m.-10:00 p.m.).

Blood tests (about 2 - 3 teaspoons) will be done once a week for a month, then once a month for 5 years, then once every 6 months (if your doctor thinks it is needed) for the remainder of your treatment on this study. A bone marrow biopsy will be done after 1-2 months of therapy to document response.

Dasatinib will be given for as long as you are responding. You will be taken off study if the disease gets worse or intolerable side effects occur.

This is an investigational study. Dasatinib is authorized for use in research only. A total of 145 patients will take part in this study. All will be treated at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >/= 18 years old who meet the following eligibility criteria
2. Patients must have one of the following hematopoietic malignancies: C-kit positive (10% or more BM or PB MNC positive by flow) acute myeloid leukemia (AML excluding acute promyelocytic leukemia) or myelodysplastic syndrome (MDS) of the following types: Refractory-relapse AML-MDS including those who fail to achieve Complete Response (CR) after the first cycle of induction; Second or subsequent AML-MDS refractory-relapse; Newly diagnosed AML-MDS patients over 60 years of age with karyotype other than t(15:17), inv16, t(8:21), who do not want chemotherapy.
3. (Con't from # 2) Patients with MDS who do not want chemotherapy as initial treatment, or who are not eligible for the treatments of higher priority.
4. Agnogenic myeloid metaplasia - myelofibrosis (MMM)
5. Hypereosinophilic syndrome (HES)
6. Polycythemia vera (PV)
7. Mastocytosis
8. Serum bilirubin less than 2mg%, serum creatinine less than 2mg% unless abnormality is considered due to hematologic malignancy by investigator.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status < 3
10. Patients must sign an informed consent indicating they are aware of the investigational nature of this study, in keeping with the policies of the hospital.
11. Women of pregnancy potential must practice an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. Prior to study enrollment, women of childbearing potential (WOCBP) (defined as not post-menopausal for 12 months or no previous surgical sterilization) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
12. Continued from #11: In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control.Women and men must continue birth control for the duration of the trial and at least 3 months after the last dose of study drug.
13. Inclusion of women and minorities: As per NIH policy, women and members of minorities will be included in this protocol as they are referred in the relevant populations. There are no exclusions of women or minorities based on the study objectives.
14. New York Heart Association (NYHA) Class < 3
15. Ph negative MPD including chronic myelomonocytic leukemia (CMML).

Exclusion Criteria:

1. Pregnant or breast-feeding women are excluded.
2. All WOCBP MUST have a negative pregnancy test prior to first receiving investigational product. If the pregnancy test is positive, the patient must not receive investigational product and must not be enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2005-11-15 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagop M Kantarjian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty-Seven participants were registered and received the study medication for this study.
Period: Overall Study
Arm/Group | Acute Myeloid Leukemia (AML) | MDS/CMML | HES/CEL | Primary Myelofibrosis (PMF) | Systemic Mastocytosis (SM)
Started | 10 | 6 | 8 | 11 | 33
Completed | 9 | 6 | 8 | 11 | 33
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acute Myeloid Leukemia (AML) | MDS/CMML | HES/CEL | Primary Myelofibrosis (PMF) | Systemic Mastocytosis (SM) | Total
Number analyzed (Participants) | 10 | 6 | 8 | 11 | 33 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5 | 8 | 28 | 46
  >=65 years | 7 | 4 | 3 | 3 | 5 | 22
Age, Continuous [Median (Full Range); unit: years] | 70 [57 to 91] | 68 [61 to 75] | 62 [23 to 75] | 63 [43 to 77] | 57 [29 to 74] | 62 [23 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 1 | 19 | 28
  Male | 7 | 4 | 5 | 10 | 14 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1
  White | 10 | 6 | 8 | 11 | 31 | 66
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 8 | 11 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: Participant Response Rate
Description: Response Rate is complete response plus partial response (CR+PR) for each disease category. Response Evaluation Criteria are as follows:
  Systemic Mastocytosis (SM): CR is the improvement of C-Findings, Tryptase <20, and no organomegaly. PR is the improvement of C-Findings.
  Acute Myeloid Leukemia (AML)/MDS and CMML: CR is bone marrow blasts </= 5%, absolute neutrophil count (ANC) >/= 1000 and platelets >/= 100. PR is bone marrow blasts 6-25% but decreased by > 50% and absolute neutrophil count, absolute neutrophil count (ANC) >/= 1000 and platelets >/= 100.
  Primary Myelofibrosis (PMF): CR is bone marrow blasts </= 5%, absolute neutrophil count (ANC) >/= 1000 and platelets >/= 100. CR is PR plus one or more of the following: ANC >/= 1000, decreased platelets by 50%, hemoglobin increase of 2g/dl or reduction splenomegaly and/or hepatomegaly by 50%.
  HES/CEL: CR is disappearance of eosinophilia </= 10%, PR is reduction of eosinophilia by >/= 50%
Time Frame: Baseline to completion of 4 week cycle or until disease progression
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Myeloid Leukemia (AML) | MDS/CMML | HES/CEL | Primary Myelofibrosis (PMF) | Systemic Mastocytosis (SM)
Number analyzed (Participants) | 9 | 6 | 8 | 11 | 33
Participants | 1 | 0 | 1 | 0 | 2

2. Secondary Outcome: Duration of Response (Survival)
Description: Response date to loss of response or last follow up.
Time Frame: Baseline, once a week for a month, thereafter monthly, up to 10 years
Population: The number of participants analyzed for duration of response reflects the number of participants with a response for each arm.
Measure: Mean (Full Range); unit: Months
Arm/Group | Acute Myeloid Leukemia (AML) | MDS/CMML | HES/CEL | Primary Myelofibrosis (PMF) | Systemic Mastocytosis (SM)
Number analyzed (Participants) | 1 | 0 | 1 | 0 | 2
Months | NA — The duration of response cannot be reported for a single participant for privacy reasons |  | NA — The duration of response cannot be reported for a single participant for privacy reasons |  | 13 [8 to 18]

ADVERSE EVENTS:
Time Frame: Through study completion, up to 10 years
Groups:
- Dasatinib All Patient Groups: Dasatinib 70 mg orally twice daily.
  Dasatinib (BMS-354825): 70 mg orally twice daily
Arm/Group | Dasatinib All Patient Groups
All-Cause Mortality (participants affected / at risk) | 2/68
Serious Adverse Events (participants affected / at risk) | 2/68
Other Adverse Events (participants affected / at risk) | 67/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib All Patient Groups (N=68)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Hemorrhage CNS (Blood and lymphatic system disorders) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib All Patient Groups (N=68)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 (18)
Edema (Blood and lymphatic system disorders) | 5 (5)
Fatigue (General disorders) | 8 (8)
Headache (General disorders) | 12 (12)
Nausea/Vomiting (Gastrointestinal disorders) | 21 (21)
Pain (General disorders) | 7 (7)
Platelets/Hemoglobin (Blood and lymphatic system disorders) | 6 (6)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
The outcome measures were collected and reported by participant diagnosis group. The Other Adverse Events and Serious Adverse Events were collected and recorded as a group for all participants registered on the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-07-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT00255346/Prot_SAP_000.pdf